CLINICAL TRIAL: NCT05797870
Title: Efficacy Evaluation of 188Re-SSS Lipiodol Selective Internal Radiation Therapy of Non Operable Hepatocellular Carcinoma Patients, a Phase II Study
Brief Title: Selective Internal Radiation Therapy and 188Re-SSS Lipiodol Treatment for Liver Cancer (Lip-Re2)
Acronym: Lip-Re2
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to the impossibility of predicting pulmonary shunts during segmental or sectoral treatment, the sponsor declared the early termination of enrolment in the trial.
Sponsor: Center Eugene Marquis (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017-1-14-010; 2020-003250-72 (EudraCT Number)
Record Dates: First submitted 2023-03-22; First posted 2023-04-04 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Hepatocellular Carcinoma Non-resectable
Keywords: Selective Internal Radiation Therapy; 188Re-SSS lipiodol
MeSH Terms: interventions — rhenium-SSS-lipiodol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 188Re-SSS lipiodol SIRT (Experimental): Patients in the experimental arm will be treated with 188Re-SSS lipiodol Selective Internal Radiotherapy (SIRT).
  Interventions: Combination Product: Selective Internal Radiation Therapy with 188Re-SSS lipiodol

INTERVENTIONS:
Combination Product: Selective Internal Radiation Therapy with 188Re-SSS lipiodol — The treatment with 188Re-SSS lipiodol SIRT requires two steps during the patient's hospitalization: the pre-treatment simulation step and the treatment step itself.
  Pre-therapeutic simulation is performed during the screening phase, before definite patient inclusion, and is composed of two procedures: a diagnostic liver angiography and a liver perfusion scintigraphy (MAA scan and SPECT/CT).
  The therapeutic stage is also composed of two procedures a therapeutic liver angiography with 188Re-SSS lipiodol and a 188Re-SSS lipiodol SPECT/CT.

SUMMARY:
The goal of this monocentric interventional study is to evaluate the efficacy, in terms of objective response rate, of the 188Re-SSS lipiodol SIRT in patients with non-operable HCC.

DETAILED DESCRIPTION:
This study is an open-labelled treatment administration study conducted with an exact one-stage one-arm study plan.

The study plans to included 35 patients and to treated 26 patients (take into account screen failures and SIRT contraindications).

The treatment is delivered by a one-day procedure leading to the injection of 188Re-SSS lipiodol. In details, the patient is hospitalized for one night. Two steps are performed while the patient is hospitalized: the pre-treatment simulation step and the treatment step itself.

After treatment, patients are followed until progression, new systemic or locoregional (in the same treatment area) antineoplastic therapy or death, within a maximum 24-month period following the SIRT.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* ECOG Performance Status 0-1
* HCC with histological diagnosis or non-invasive diagnosis according to AASLD criteria
* Non operable and not accessible to ablation therapy
* At least one measurable lesion using mRECIST
* Tumor involvement <50% of the liver
* BCLC classification A to C
* Compensated cirrhosis (Child Pugh A or B7), if cirrhosis present
* Registration with a social security scheme
* Written and informed consent of the patient or his/her legal representative

Exclusion Criteria:

* Inadequate hematological, hepatic, renal, thyroid and coagulation functions:

  1. Hemoglobin < 8,5 g/dl
  2. Granulocytes < 1500/mm3
  3. Platelets< 50 000 /mm3
  4. Bilirubin level ≥ 35 mol/l
  5. Transaminases > 6 UNL
  6. Creatinine > 1,5 UNL
  7. TSH < 0,2 µUI/L
* Chronic respiratory insufficiency history
* Known hemophilia with exophytic tumor > 1 cm
* Extra-hepatic metastasis except hilum node < 2 cm
* Lung shunt >20% evaluated with 99mTc albumin macroaggregate (MAA)
* Poor tumor targeting with 99mTc albumin macroaggregate (MAA)
* Previous SIRT
* Previous systemic treatment within 4 weeks before radioembolization
* More than 2 previous TACE (or embolization), in the area to be treated
* Other neoplasia except if complete remission from at least one year
* Contraindication related to the technique, in particular severe arterial pathology of the lower limbs or the aorta contraindicating or making difficult an arteriography by femoral approach
* Pregnant woman or likely to be or breastfeeding, or male or female patients of reproductive potential without effective contraception from screening to 1 month after the end of the treatment
* Minors, individual deprived of liberty, or under any kind of guardianship or trusteeship.
* Patients unable to submit to medical follow-up of the study for social, medical or psychological reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2024-02-14 (Actual); Primary Completion 2025-12-14 (Estimated); Study Completion 2027-02-26 (Estimated)

PRIMARY OUTCOMES:
The objective response rate | through study completion, an average of 4 year
  Defined as the best overall response occurring within 6 months' post 188Re-SSS lipiodol injection according to the modified RECIST criteria for hepatocellular carcinoma

CONTACTS AND LOCATIONS:
Overall Officials: Etienne Garin, MD PHD, Principal Investigator — Centre de Lutte contre le Cancer Eugène Marquis
Locations (1):
- Centre de Lutte contre le Cancer Eugène Marquis, Rennes, Brittany Region, France